CLINICAL TRIAL: NCT04459195
Title: An Investigation of Acute Effects of Static Stretching Duration on Gastrocnemius Muscle Vascularization by Superb Microvascular Imaging Method
Brief Title: Acute Effects of Static Stretching Duration on Gastrocnemius Muscle Vascularization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Kamile UZUN AKKAYA, Principal Investigator, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kamile U Akkaya
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-12

CONDITIONS: Muscle Stretching Exercises
Keywords: Gastrocnemius; Static Stretching; Muscle Vascularization; Superb Microvascular Imaging
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2 Minute Static stretching (Experimental): Stretching applications will be applied to the first group for 2 minutes .
  Interventions: Behavioral: 2 Minute Static Stretching
- 5 Minute Static stretching (Experimental): Stretching applications will be applied to the first group for 5 minutes.
  Interventions: Behavioral: 5 Minute Static Stretching

INTERVENTIONS:
Behavioral: 2 Minute Static Stretching — Stretching applications will be applied to the first group for 2 minutes. Static stretching exercise will be performed under the supervision of a physiotherapist as 30 seconds of stretching and 30 seconds of rest and and the individuals will be asked to participate in the exercise actively.
  Arms: 2 Minute Static stretching
Behavioral: 5 Minute Static Stretching — Stretching applications will be applied to the first group for 5 minutes. Static stretching exercise will be performed under the supervision of a physiotherapist as 30 seconds of stretching and 30 seconds of rest and and the individuals will be asked to participate in the exercise actively.
  Arms: 5 Minute Static stretching

SUMMARY:
Stretching effects skeletal muscle flexibility, vascularity and physical performance. The aim of our study is to examine the acute effects of static stretching duration on gastrocnemius muscle vascularization in healthy participants by superb microvascular imaging (SMI) and to compare the effects of 2 and 5 minutes of static stretching on blood flow.

DETAILED DESCRIPTION:
The study will be included 30 healthy volunteers. The participants will be divided into two groups. Static stretching was administered to the gastrocnemius muscle. Stretching applications will be applied to the first group for 2 minutes and to the second group for 5 minutes. Muscle vascularization will be evaluated by a new method, superb microvascular imaging (SMI). SMI is a recently developed ultrasound imaging technique that aims to visualize low velocity and small diameter blood vessel flow.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers between the ages of 18-35,
* Without knee, hip, ankle and waist pathology,
* Has not undergone any surgery on the lower extremity.

Exclusion Criteria:

* Rheumatic, musculoskeletal, neurological and vestibular problems,
* Bone pathologies,
* Joint laxity,
* Connective tissue disorders
* Diabetes, metabolic syndrome, arthritic or inflammatory problems

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Muscle vascularization | Immediately after the application.
  The evaluation of muscle vascularization will be made using the Superb microvascular imaging method by a radiologist. Superb microvascular imaging is a recently developed ultrasound imaging technique that aims to visualize low velocity and small diameter blood vessel flow.
Muscle vascularization | 10 minutes after the application.
  The evaluation of muscle vascularization will be made using the Superb microvascular imaging method by a radiologist. Superb microvascular imaging is a recently developed ultrasound imaging technique that aims to visualize low velocity and small diameter blood vessel flow.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Caliskan E, Akkoc O, Bayramoglu Z, Gozubuyuk OB, Kural D, Azamat S, Adaletli I. Effects of static stretching duration on muscle stiffness and blood flow in the rectus femoris in adolescents. Med Ultrason. 2019 May 2;21(2):136-143. doi: 10.11152/mu-1859. PMID 31063516
- [Background] Maeda N, Urabe Y, Tsutsumi S, Sakai S, Fujishita H, Kobayashi T, Asaeda M, Hirata K, Mikami Y, Kimura H. The Acute Effects of Static and Cyclic Stretching on Muscle Stiffness and Hardness of Medial Gastrocnemius Muscle. J Sports Sci Med. 2017 Dec 1;16(4):514-520. eCollection 2017 Dec. PMID 29238251
- [Background] Nakamura M, Ikezoe T, Nishishita S, Umehara J, Kimura M, Ichihashi N. Acute effects of static stretching on the shear elastic moduli of the medial and lateral gastrocnemius muscles in young and elderly women. Musculoskelet Sci Pract. 2017 Dec;32:98-103. doi: 10.1016/j.msksp.2017.09.006. Epub 2017 Sep 25. PMID 28988152
- [Background] Jiang ZZ, Huang YH, Shen HL, Liu XT. Clinical Applications of Superb Microvascular Imaging in the Liver, Breast, Thyroid, Skeletal Muscle, and Carotid Plaques. J Ultrasound Med. 2019 Nov;38(11):2811-2820. doi: 10.1002/jum.15008. Epub 2019 Apr 5. PMID 30953387